CLINICAL TRIAL: NCT06827210
Title: Treatment of Bulbar Urethral Strictures With Optilume Drug-Coated Balloons in an Untreated Population
Acronym: FIRST-CARE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Gødstrup Hospital (Other); Regionshospital Nordjylland (Other Government)
Responsible Party: Principal Investigator, Marco Bassam Mahdi, MD, PhD Fellow, Principal Investigator, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F2024-214
Record Dates: First submitted 2025-01-30; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Urethral Stricture; Urethral Stricture, Anterior; Urethral Stricture, Male; Urethral Stricture Less Than 2 cm
Keywords: Urethral Stricture; Optilume Drug-Coated Balloon; DVIU; Urology; Patient-Reported Outcomes
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Optilume Drug-Coated Balloon (DCB) (Experimental): Participants in this arm will receive treatment with the Optilume drug-coated balloon (DCB), which combines mechanical dilation with localized drug delivery of paclitaxel to reduce stricture recurrence and promote healing.
  Interventions: Device: Optilume DCB
- Standard Direct Visual Internal Urethrotomy (DVIU) (Active Comparator): Participants in this arm will undergo standard Direct Visual Internal Urethrotomy (DVIU), a commonly performed endoscopic procedure for the treatment of bulbar urethral strictures.
  Interventions: Procedure: Standard Direct Visual Internal Urethrotomy (DVIU)

INTERVENTIONS:
Device: Optilume DCB — Optilume DCB is a drug-coated balloon catheter designed for the treatment of bulbar urethral strictures. It combines mechanical dilation with localized drug delivery to reduce stricture recurrence and promote urethral healing. The balloon is coated with paclitaxel, an antiproliferative agent, to minimize scar tissue formation and improve treatment outcomes.
  Other Names: Drug-coated balloon
  Arms: Optilume Drug-Coated Balloon (DCB)
Procedure: Standard Direct Visual Internal Urethrotomy (DVIU) — Standard Direct Visual Internal Urethrotomy (DVIU), also known as Sachse Internal Urethrotomy, is a minimally invasive endoscopic procedure for treating urethral strictures.
  Other Names: Sachse Internal Urethrotomy
  Arms: Standard Direct Visual Internal Urethrotomy (DVIU)

SUMMARY:
This randomized controlled trial investigates the effectiveness and safety of the Optilume® drug-coated balloon (DCB) compared to standard direct visual internal urethrotomy (DVIU) in the treatment of bulbar urethral strictures. The primary objective is to assess freedom from repeat intervention at 12 months. Secondary objectives include evaluating urethral patency, urinary symptoms, and sexual function through objective measures (Qmax, PVR, cystoscopy) and patient-reported outcomes (USS-PROM, IPSS, IIEF-5). The study will recruit 140 participants across multiple sites, with follow-ups conducted at 6 and 12 months. This trial seeks to provide evidence for Optilume DCB as a safe and effective alternative to standard treatment.

DETAILED DESCRIPTION:
This randomized controlled trial aims to evaluate the safety and efficacy of the Optilume® drug-coated balloon (DCB) in the treatment of bulbar urethral strictures. The trial includes adult male participants who have not received prior treatment for urethral strictures. Participants will be randomly assigned to one of two treatment groups: Optilume DCB or standard direct visual internal urethrotomy (DVIU).

The primary objective of the study is to compare the recurrence rate of urethral strictures at 12 months between the two groups. Secondary objectives include assessing patient-reported outcomes (using USS-PROM, IPSS, and IIEF-5), urethral patency (via Qmax and post-void residual volume), and safety (monitoring adverse events).

Follow-Up Schedule:

At Diagnosis: Baseline assessments will include cystoscopy, uroflowmetry (Qmax), post-void residual (PVR), patient-reported outcomes (USS-PROM, IPSS, and IIEF-5), and demographic data (age, sex, BMI, comorbidities, and smoking status). Informed consent will also be obtained.

Day 3 (Foley Removal): Participants will return for catheter removal. 6-Month Follow-Up: Assessments will include Qmax, PVR, and patient-reported outcomes (USS-PROM, IPSS, and IIEF-5).

12-Month Follow-Up: Final assessments will include cystoscopy, Qmax, PVR, and patient-reported outcomes (USS-PROM, IPSS, and IIEF-5).

The study will recruit 140 participants across multiple sites, with recruitment anticipated to span approximately 17.5 months. Data will be analyzed using Kaplan-Meier survival curves to compare recurrence rates, and log-rank tests will be used to assess statistical significance. Modified Poisson regression will be applied to evaluate potential confounders.

This study aims to provide robust evidence on the effectiveness of Optilume DCB in reducing stricture recurrence, improving patient outcomes, and offering a safe alternative to standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 18 years or older.
* Diagnosed with a treatment-naive, single bulbar urethral stricture.
* Stricture length ≤3 cm.
* Eligible for local treatment with paclitaxel.
* Able to provide written informed consent.

Exclusion Criteria:

* Female (chromosomal) sex.
* History of prior urethral stricture or prior treatment thereof.
* History of hypospadias repair.
* History of genital lichen sclerosis.
* Active or unresolved confounding etiology, including bladder neck contracture, neurogenic bladder, known or being evaluated for symptomatic benign prostatic hyperplasia (BPH) or surgical treatment for BPH within the last 5 years.
* Known allergy or hypersensitivity to paclitaxel or any component of the Optilume DCB.
* Known peripheral artery disease.
* Severe comorbidities with an American Society of Anesthesiologists (ASA) score of 4 or higher.
* Patients unable to comply with follow-up protocols or provide informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-02-07 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Freedom from Repeat Intervention at 12 Months | 12 months post-intervention
  "The primary outcome is the proportion of participants who remain free from repeat intervention for urethral stricture recurrence at 12 months following treatment. Repeat intervention is defined as any procedure to address stricture recurrence, such as dilation, DVIU, or urethroplasty. Referrals for repeat interventions made within the 12-month follow-up period will also be included, even if the procedure itself is scheduled beyond the 12-month mark."

SECONDARY OUTCOMES:
Urethral Patency Assessed via Cystoscopy at 12 Months | 12 months post-treatment
  Urethral patency will be assessed using cystoscopy at 12 months. Patency is defined as the absence of visually confirmed narrowing that compromises the urethral lumen.
Maximum Urinary Flow Rate (Qmax) at 12 Months | 12 months post-treatment
  The maximum urinary flow rate (Qmax) will be measured using uroflowmetry at 12 months as an indicator of urethral function. An improvement in Qmax is considered indicative of treatment success.
Post-Void Residual (PVR) Volume at 12 Months | 12 months post-treatment
  Post-void residual (PVR) volume will be assessed using ultrasound at 12 months to evaluate bladder emptying efficiency. Lower PVR values are associated with successful treatment outcomes.
Urethral Stricture Surgery Patient-Reported Outcome Measure (USS-PROM) | 12 months post-treatment
  The Urethral Stricture Surgery Patient-Reported Outcome Measure (USS-PROM) is a patient-reported outcome measure consisting of: (1) Lower Urinary Tract Symptoms Construct (Q1-6) from International Consultation on Incontinence Questionnaire Male Lower Urinary Tract Symptoms Module (0-24, higher = worse symptoms); (2) LUTS-Specific QoL (Q7) (1-4, higher = worse QoL); (3) Peeling's Voiding Picture (Q8) (1-4, 1 = worst, 4 = best voiding); and (4) EQ-5D with an index value (1.000 to 0.033, higher = better health) and EQ-Visual Analogue Scale (0-100, higher = better health status), based on the Danish EQ-5D-5L Value Set (PMID 33527304).
International Prostate Symptom Score (IPSS) at 12 Months | 12 months post-treatment
  The International Prostate Symptom Score (IPSS) is a patient-reported outcome measure assessing lower urinary tract symptoms (LUTS). It consists of seven symptom questions (Q1-7) scored from 0 to 5 (0 = no symptoms, 5 = most severe), with a total score range of 0 to 35 (higher = worse symptoms). An additional Quality of Life (QoL) question (Q8) is scored from 0 to 6 (0 = delighted, 6 = terrible), assessing the patient's perception of urinary symptoms.
International Index of Erectile Function (IIEF-5) at 12 Months | 12 months post-treatment
  The International Index of Erectile Function-5 (IIEF-5) is a patient-reported outcome measure assessing erectile function. It consists of five questions (Q1-5), each scored from 1 to 5, with a total score range of 5 to 25. Higher scores indicate better erectile function, while lower scores suggest increasing severity of erectile dysfunction (22-25 = no dysfunction, 17-21 = mild, 12-16 = mild-moderate, 8-11 = moderate, 5-7 = severe).
Incidence of Adverse Events (AEs) | From enrollment to 12 months post-treatment
  The incidence of adverse events (AEs) related to the intervention will be documented throughout the study. AEs include any unexpected or undesirable events, categorized by severity and relationship to the treatment.
Incidence of Postoperative Complications | 12 months post-treatment
  The incidence of postoperative complications will be documented and categorized based on their severity.

CONTACTS AND LOCATIONS:
Overall Officials: Tommy K Nielsen, MD, PHD, Principal Investigator — Aalborg University Hospital; Marco B Mahdi, MD, Principal Investigator — Aalborg University Hopsital; Henrik Weinreich, MD, Principal Investigator — Regionshospital Nordjylland; Charlotte H Graugaard-Jensen, MD, PHD, Principal Investigator — Gødstrup Hospital
Locations (3):
- Denmark (3):
  - Gødstrup Regional Hospital, Gødstrup, Central Jutland
  - Aalborg University Hospital, Aalborg, Region North Jutland
  - North Denmark Regional Hospital, Hjørring, Region North Jutland

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data (IPD) will be shared upon reasonable request submitted to the sponsor and evaluated by the steering committee. Researchers must submit a formal request detailing the intended use. Approval will require signing a data access agreement to ensure the data is only used for predefined and accepted research purposes.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after the study's primary completion date and will be accessible for a period of 5 years.
Access Criteria: Researchers requesting access must submit a formal request to the sponsor, outlining the intended use of the data. Access will be granted upon approval by the steering committee and will require signing a data access agreement to ensure responsible use.

REFERENCES:
- [Result] Al Taweel W, Seyam R. Visual Internal Urethrotomy for Adult Male Urethral Stricture Has Poor Long-Term Results. Adv Urol. 2015;2015:656459. doi: 10.1155/2015/656459. Epub 2015 Oct 1. PMID 26494995
- [Result] Harraz AM, El-Assmy A, Mahmoud O, Elbakry AA, Tharwat M, Omar H, Farg H, Laymon M, Mosbah A. Is there a way to predict failure after direct vision internal urethrotomy for single and short bulbar urethral strictures? Arab J Urol. 2015 Dec;13(4):277-81. doi: 10.1016/j.aju.2015.07.007. Epub 2015 Sep 3. PMID 26609447
- [Result] Redon-Galvez L, Molina-Escudero R, Alvarez-Ardura M, Otaola-Arca H, Alarcon Parra RO, Paez-Borda A. Predictors of urethral stricture recurrence after endoscopic urethrotomy. Actas Urol Esp. 2016 Oct;40(8):529-33. doi: 10.1016/j.acuro.2016.03.013. Epub 2016 May 17. English, Spanish. PMID 27207599
- [Result] Elliott SP, Coutinho K, Robertson KJ, D'Anna R, Chevli K, Carrier S, Aube-Peterkin M, Cantrill CH, Ehlert MJ, Te AE, Dann J, DeLong JM, Brandes SB, Hagedorn JC, Levin R, Schlaifer A, DeSouza E, DiMarco D, Erickson BA, Natale R, Husmann DA, Morey A, Olsson C, Virasoro R. One-Year Results for the ROBUST III Randomized Controlled Trial Evaluating the Optilume(R) Drug-Coated Balloon for Anterior Urethral Strictures. J Urol. 2022 Apr;207(4):866-875. doi: 10.1097/JU.0000000000002346. Epub 2021 Dec 2. PMID 34854748
- [Result] Virasoro R, DeLong JM, Estrella RE, Pichardo M, Rodriguez Lay R, Espino G, Elliott SP. A Drug-Coated Balloon Treatment for Urethral Stricture Disease: Three-Year Results from the ROBUST I Study. Res Rep Urol. 2022 May 6;14:177-183. doi: 10.2147/RRU.S359872. eCollection 2022. PMID 35572815
- [Result] Barbagli G, Fossati N, Montorsi F, Balo S, Rimondi C, Larcher A, Sansalone S, Butnaru D, Lazzeri M. Focus on Internal Urethrotomy as Primary Treatment for Untreated Bulbar Urethral Strictures: Results from a Multivariable Analysis. Eur Urol Focus. 2020 Jan 15;6(1):164-169. doi: 10.1016/j.euf.2018.10.014. Epub 2018 Nov 6. PMID 30409684
- [Result] Kluth LA, Ernst L, Vetterlein MW, Meyer CP, Reiss CP, Fisch M, Rosenbaum CM. Direct Vision Internal Urethrotomy for Short Anterior Urethral Strictures and Beyond: Success Rates, Predictors of Treatment Failure, and Recurrence Management. Urology. 2017 Aug;106:210-215. doi: 10.1016/j.urology.2017.04.037. Epub 2017 May 4. PMID 28479479
- [Derived] Mahdi MB, Haase RN, Sander L, Tuckus G, Liltorp DL, Jorgensen L, Graugaard-Jensen CH, Weinreich H, Pennisi CP, Nielsen TK. Treatment of bulbar urethral strictures with Optilume drug-coated balloons in a previously untreated population (FIRST-CARE): protocol for a single-blind multicentre randomised controlled trial. BMJ Open. 2026 Jan 8;16(1):e103948. doi: 10.1136/bmjopen-2025-103948. PMID 41506760